CLINICAL TRIAL: NCT06594926
Title: Evaluating the Efficacy of Bipolar Androgen Therapy in Extending Metastasis-free Survival in Patients With M0 Castrate-resistant Prostate Cancer With PSA Progression But Not Radiological or Clinical Progression on Darolutamide
Brief Title: Working Out M0 Bipolar Androgen Therapy
Acronym: WOMBAT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Australian and New Zealand Urogenital and Prostate Cancer Trials Group (Other)
Collaborators: Bayer (Industry); The George Institute (Other); HMRI (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANZUP 2201
Record Dates: First submitted 2024-05-23; First posted 2024-09-19 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
Keywords: darolutamide; testosterone; bipolar androgen therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — testosterone enanthate

STUDY DESIGN:
Intervention Model Description: This is a single-arm phase 2 prospective, interventional study to assess the efficacy and safety of cyclical testosterone and darolutamide in non-metastatic castration-resistant prostate cancer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Testosterone enthanate (Experimental): Participants will receive continuous androgen deprivation therapy with LHRH agonists/antagonists. The study intervention will be IM testosterone enthanate, injected on day 1 of each 56-day cycle (+3 days) except for cycle 1. Concurrent darolutamide will be taken at a dose of 600mg BD on days 29-56 of each cycle. Both LHRH and agonist/antagonist and darolutamide are supplied through the PBS as standard of care medications.
  Interventions: Drug: Testosterone Enanthate

INTERVENTIONS:
Drug: Testosterone Enanthate — Testosterone enanthate is a depot formulation used in Australia typically for androgen replacement in people with confirmed testosterone deficiency.
  Other Names: Primoteston Depot

SUMMARY:
The WOMBAT study will test if BAT can prolong the time it takes for nmCRPC prostate cancer to become detectable in other areas of the body (metastatic disease).

Approximately 69 participants over the age of 18 with castrate resistant prostate cancer, no evidence of metastatic disease (M0) on conventional imaging (WBBS and CT scan at screening) and PSA only progression on darolutamide will be enrolled from approximately 8 sites within Australia.

Participants will receive continuous androgen deprivation therapy with LHRH agonists/antagonists. The study intervention will be IM testosterone enthanate, injected on day 1 of each 56-day cycle. Concurrent darolutamide will be taken at a dose of 600mg BD on days 29-56 of each cycle. Both LHRH and agonist/antagonist and darolutamide are supplied through the PBS as standard of care medications. Administration of both testosterone and darolutamide will continue until disease progression, beyond disease progression, unacceptable toxicity, death, withdrawal of consent or study Sponsor termination of the study.

Primary objective (endpoint) is to determine the metastasis-free survival (time from commencing BAT to evidence of metastases or death)

DETAILED DESCRIPTION:
This is a study to assess the efficacy and safety of cyclical testosterone and darolutamide in non-metastatic castration-resistant prostate cancer.

Adults with castrate resistant prostate cancer, with no evidence of metastatic disease (M0) on conventional imaging [Whole Body Bone Scan (WBBS) and Computed Tomography (CT) scan at screening] and prostate specific antigen (PSA) only progression on darolutamide may be eligible.

Study participants will receive cyclical treatment with intramuscular (IM) testosterone, darolutamide and ongoing medical/surgical castration. This will be delivered in 56-day cycles until evidence of metastatic disease on conventional imaging unless treated beyond progression. Participants will be asked to provide blood samples, complete questionnaires and undergo scans during their treatment.

It is hoped that findings from this study will help develop new treatment pathways for those with non-metastatic castration-resistant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the prostate
2. ≥18 years of age
3. ECOG performance status 0-1
4. PSA progression while on darolutamide defined as three rising PSA (1 baseline and 2 consecutive rises) levels at least 1 week apart despite castrate testosterone level (<1.7nmol/L). Patients with a minor subsequent PSA fall, provided there was no intervening therapy since the three consecutive rises, are eligible
5. AJCC stage M0 on conventional imaging.

   1. Previous PSMA PET only M1 disease in the hormone-sensitive setting that is now M0 CRPC on conventional imaging following >18 months of ADT + darolutamide are eligible.
   2. Nodes up to 2cm in short-axis in pelvis are permitted
6. PSA >1.0 ng/mL during screening
7. Serum testosterone <1.7nmol/L and on an LHRH agonist/antagonist
8. Adequate bone marrow function (platelets > 100 x 109/L, ANC > 1.5 x 109/L, Hb >90)
9. Adequate liver function (ALT or AST < 2.5 x ULN, bilirubin < 1.5 x ULN)
10. Adequate renal function (creatinine <1.5 x ULN)
11. Willingness and ability to comply with study requirements, including treatment and timing of treatment.

Exclusion Criteria:

1. Life expectancy <3 months.
2. Neuroendocrine or small cell prostate cancer on any prior diagnostic tissue sample.
3. Metastatic prostate cancer on conventional imaging (WBBS or CT scan) at any point in disease course (except for pathological nodes up to 2cm in short axis in the pelvis).
4. Current or prior treatment with enzalutamide, abiraterone, apalutamide, or cytotoxic chemotherapy. Patients with pelvic nodal metastases (below the aortic bifurcation) <2cm in short axis at original diagnosis who ceased cytotoxic chemotherapy (docetaxel) at least 12 months prior to C1D1 are eligible. Prior first generation ARSI such as bicalutamide, flutamide, nilutamide are permitted.
5. Current or pre-existing cardiac or thromboembolic risk factors, including but not limited to:

   i. Prior myocardial infarction, or unstable angina within 24 months of study entry, ii. Uncontrolled or symptomatic cardiac disease including, but not limited to angina, dyspnoea on exertion, orthopnoea; cardiac failure (NYHA classification 3-4) or uncontrolled arrhythmias.

   iii. Significant co-morbidities that increase cardiovascular risk, including significant hypertension (Baseline systolic BP>160 or diastolic BP>100 despite optimal treatment) that are uncontrolled, as assessed by the treating oncologist.
6. Another malignancy diagnosis within 2 years before registration. Participants with a history of treated carcinoma in situ, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or non-muscle invasive urothelial carcinoma of the bladder are eligible if malignancy has been treated with curative intent. Participants with a history of other malignancies are eligible if they have been continuously disease-free for at least 2 years after definitive primary treatment or the chance of recurrence is sufficiently low as to be very unlikely to affect study outcomes according to the treating local oncologist.
7. Concurrent illness that could preclude the participant's ability to participate in the study and follow protocol with reasonable safety.
8. Planned ongoing drug Interactions as per protocol section 5.2.4 that are considered unable to be managed prior to study registration.
9. Radiation therapy within the previous 4 weeks (participants are permitted to have SBRT to PSMA PET only disease prior to study enrolment if they continue on darolutamide. Note that if the metastases are visible on conventional imaging at the time of radiation treatment the participant is not eligible).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Metastases free survival | From date of commencing Bipolar Androgen Therapy (BAT) until first documented evidence of metastatic disease or date of death, assessed every 8 weeks, on average 4 years
  Based on PCWG3 criteria (appendix 2) and/or RECIST1.1 (appendix 1) on CT and WBBS imaging.

SECONDARY OUTCOMES:
Safety and tolerability of BAT + darolutamide | Continuously throughout the study, from time of commencing BAT until 30 days after last dose of treatment
  The safety and tolerability of BAT + darolutamide (Incidence and grade of AEs by NCI CTCAE v5.0 Common Terminology Criteria for Adverse Events will be used to grade and classify adverse events after each cycle. Adverse events will be reported as all grade, grade 3-4, grade 5 and Adverse events of special interest (related to bipolar androgen therapy).
The effect of BAT + darolutamide on Health-related Quality of Life QLQ-C30 | During screening and then every 2 weeks upon commencement of BAT for 8 weeks and then every 4 weeks until last dose of treatment, on average 2 years.
  Using the European Organisation for Research Treatment of Cancer (EORTC) quality of life (QOL) questionnaire QLQ-C30. QLQ-C30 uses 28 questions about overall QOL with each question answerable using a scale from 1 (not at all) to 4 (very much). Overall scores can be from a minimum of 28 indicating a better QOL and higher scores with a maximum of 112 indicating lower overall QOL. It has two summary questions which asks participants to rank, 1) overall health and 2) overall QOL on scale from 1: very poor, to 7; excellent.
The effect of BAT + darolutamide on Health-related Quality of Life QLQ-PR25 | During screening and then every 2 weeks upon commencement of BAT for 8 weeks and then every 4 weeks until last dose of treatment, on average 2 years.
  Using the European Organisation for Research Treatment of Cancer (EORTC) quality of life (QOL) questionnaire QLQ-PR25. QLQ-PR25 is a supplement to QLQ-C30 and designed to assess symptoms related to prostate cancer, treatment, and aspects of life related to prostate cancer.QLQ-PR25 uses 25 questions about overall QOL with each question answerable using a scale from 1 (not at all) to 4 (very much). Overall scores can be from a minimum of 25 indicating a better QOL and higher scores with a maximum of 100 indicating lower overall QOL.
PSA response rate to BAT + darolutamide | During screening and then every 2 weeks from the time of commencing BAT for first 8 weeks and then every 4 weeks until last dose of treatment, on average 2 years
  By testing PSA level in blood. PSA response rate is defined as a PSA reduction of >=50% from baseline as per PCWG3 criteria
Time to PSA progression on BAT + darolutamide | During screening and then every 2 weeks from the time of commencing BAT for first 8 weeks and then every 4 weeks until last dose of treatment, on average 2 years
  By testing PSA level in blood. PSA progression is defined as a PSA increase of >=25% from baseline or nadir, confirmed on subsequent test >=1 week later as per PCWG3)
PSA and hormone kinetics in response to BAT + darolutamide. This will be assessed as a composite outcome. | Every 2 weeks for first 24 weeks from the time of commencing BAT
  Blood tests assessing change in PSA, testosterone, oestradiol, Dihydrotestosterone (DHT), Dehydroepiandrosterone (DHEA), sex hormone-binding globulin (SBHG)
The effect of BAT + darolutamide on metabolic and bone turnover markers and bone mineral density. This will be assessed as a composite outcome. | Serum/plasma/urine - at screening and at 6 and 12 months on treatment. Bone densitometry imaging - at screening and 12 months on treatment.
  Testing bone turnover markers via serum procollagen type I N propeptide (PINP) and plasma C-terminal cross-linking telopeptide of type I collagen (CTX). Bone densitometry imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Joshua, Study Chair — St Vincent's Hospital, Sydney
Locations (12):
- Australia (12):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - The Border Cancer Hospital, Albury, New South Wales
  - St Vincents Hospital, Darlinghurst, New South Wales
  - GenesisCare North Shore, St Leonards, New South Wales
  - Sydney Adventist Hospital, Wahroonga, New South Wales
  - ICON Cancer Centre, Chermside, Queensland
  - Mater Misericordiae Ltd - QLD, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Grampians Health, Ballarat, Victoria
  - Eastern Health - Box Hill, Box Hill, Victoria
  - Cabrini Health, Malvern, Victoria
  - Northeast Health Wangaratta, Wangaratta, Victoria

IPD SHARING:
Plan to Share IPD: No